CLINICAL TRIAL: NCT06003608
Title: Observational, Cross-sectional Clinical Study in Parkinson's Disease (PD) Patients and Healthy Controls (HC) to Identify PD Specific Microbial and Metabolic Fingerprints in Small Intestinal (SI) Fluid and Blood
Brief Title: Observational Small Intestine and Blood Fingerprint (SmIle) Study in Parkinson's Disease
Acronym: SmIle
Status: Active, not recruiting | Type: Observational
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: MRM Health NV (Industry)
Responsible Party: Sponsor
Other Study IDs: M007-PD-001
Record Dates: First submitted 2023-08-02; First posted 2023-08-22 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood sample, Stool sample, Fluid from small intestine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy control (HC): 25 neurotypical controls, age-matched to the Parkinson's disease group
  Interventions: Device: Fluid biopsy capsule
- Parkinson's disease (PD): 75 Parkinson's disease patients
  Interventions: Device: Fluid biopsy capsule; Drug: Levodopa-Carbidopa Immediate Release

INTERVENTIONS:
Device: Fluid biopsy capsule — Ingestion of two SIMBA capsules
Drug: Levodopa-Carbidopa Immediate Release — Single dose, Levodopa-Carbidopa Immediate Release
  Groups: Parkinson's disease (PD)

SUMMARY:
Observational cross-sectional study in PD patients and healthy controls (HC) using an investigational medical device consisting of a passive small intestine microbiome aspiration (SIMBA) system (capsule) that is ingested orally and recovered together with the stools (home recovery) together with blood sampling (during the onsite visit).

DETAILED DESCRIPTION:
Participants will be swallowing two SIMBA capsules which allows for minimally-invasive sampling of the microbiome and metabolome deep in the small intestine. Researchers will use the capsule samples to determine the small intestinal microbiome and metabolomic signatures in luminal fluid samples from the small bowel in Parkinson Disease (PD) patients compared to healthy controls (HC).

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to be included in the study only if all of the following criteria apply:

1. Males and females aged 50-85 years old at time of on-site visit
2. Signed Informed consent
3. Willing & able to comply with study procedures (including SIMBA capsule ingestion) and have study assessments performed
4. Able to swallow a size-00 capsule (23mm length) in OFF state Additional inclusion criteria for PD patients only
5. Diagnosis of idiopathic PD (Clinically Probable PD), including documented levodopa responsiveness
6. Treatment with an immediate release levodopa formulation during the day at a stable dose for at least 2 months prior to enrollment

Exclusion Criteria

Subjects are excluded from the study if any of the following criteria apply:

1. Any risk of capsule non-excretion, including, e.g., prior gastrointestinal disease, surgery, or radiation treatment which, in the Investigator's opinion, would lead to intestinal structuring or obstruction, achalasia, eosinophilic esophagitis, any inflammatory bowel disease (IBD), cancer diagnosis or treatment within the past year, or previous esophageal, gastric, small intestinal, or colonic surgery; appendectomy or cholecystectomy more than 3 months prior to on-site study visit are acceptable,
2. Use of any medications in the week prior to the on-site study visit, unless part of regular treatment, that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics); laxative use is allowed provided that it is kept unchanged in the week prior to the study visit. PPIs are allowed provided a wash-out period of 48 hours is respected before swallowing the SIMBA capsules and PPI treatment is resumed only 4 hours thereafter,
3. Any contraindication for using domperidone, including a long QT interval, concomitant use of QT prolonging drugs, any risk of significant electrolyte abnormality, known hypersensitivity, known liver impairment or significant (e.g. unstable) cardiac disease (see label) putting the subject at significant risk according to the investigator's clinical judgement
4. History of oropharyngeal dysphagia, or other swallowing disorder with a risk of capsule aspiration, e.g. SDQ score > 4,
5. Any concomitant PD treatment, including any dopamine agonist and MAO-B inhibitor, except (for PD patients only) an immediate release levodopa formulation during the day (required per inclusion criterion), the concomitant use of a decarboxylase inhibitor and the use of a controlled release levodopa formulation at bedtime,
6. Major genital and/or rectum prolapse,
7. Any concomitant or previous treatment (<2 months from on-site study visit) with significant anti-inflammatory or immune suppressant medication, e.g. DMARDs, biologicals or systemic corticosteroids, except non-chronic PRN use of an NSAID and/or 5-ASA (mesalazine) treatment,
8. Active cancer, including any prolactinoma, within 5 years (allowed: uncomplicated basal cell carcinoma and successfully removed carcinoma in situ),
9. Clinically significant immune deficiency (according to Investigator's judgement),
10. Documented HIV infection, or any clinically significant systemic infection,
11. Antibiotic use (except for local use), use of prebiotics, or probiotics ≤12 weeks prior to on-site study visit, or Fecal Microbiota Transplantation anytime in medical history
12. Dementia in medical history or identified by a MMSE <24,
13. Insulin-dependent diabetes mellitus,
14. Current Psychosis episode by clinical judgement based on anamnesis
15. Active significant impulse control disorder (by clinical judgement and based on interview and medical records)
16. Pregnancy
17. Alcohol or drug abuse
18. Deep brain stimulation or Duodopa/Lecigon treatment.
19. Subject, according to investigator assessment, not expected to be able to comply with study procedures including SIMBA capsule recovery and SIBO breath test execution with - or without help (when home).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligibility will be determined based on information reported by the subject and the results of the screening assessments (physical exam, etc). Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Difference in microbiome profile of small intestine samples between groups | Baseline
  Functional dysbiosis profile of the small intestinal microbiota of Parkinson's Disease patients compared to age-matched neurotypical controls, as determined by whole metagenome shotgun sequencing based profiling

SECONDARY OUTCOMES:
Difference in blood metabolome composition between groups | Baseline
  Blood metabolome composition profile of Parkinson's Disease patients as compared to age-matched neurotypical controls, as determined by metabolomics analysis
Correlation between the observed small intestine microbiome profile and blood metabolome composition, including, in PD subjects, levodopa pharmacodynamics | Baseline
  Small intestinal and blood pharmacodynamics of Levodopa as a function of small intestinal microbiota profiles, as determined by blood and small intestinal metabolomics and small intestinal whole metagenome shotgun profiling and appropriate statistical correlation methods

CONTACTS AND LOCATIONS:
Overall Officials: Davide Martino, MD PHD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No